CLINICAL TRIAL: NCT03968315
Title: Can MRI Replace CT in the Evaluation of Thymoma?
Brief Title: An Investigational Scan (MRI) in Imaging Patients With Newly-Diagnosed or Recurrent Thymoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 2011-0360; NCI-2019-02643 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0360 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Malignant Thymoma; Thymoma
MeSH Terms: conditions — Thymoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (MRI, diaphragm fluoroscopy) (Experimental): Patients undergo an MRI scan over 45-60 minutes and a diaphragm fluoroscopy 30 days before surgery.
  Interventions: Procedure: Diaphragm Fluoroscopy; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Diaphragm Fluoroscopy — Undergo diaphragm fluoroscopy
  Other Names: Sniff Test
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This trial studies the accuracy of a magnetic resonance imaging (MRI) scan in imaging the inside of the chest in patients with thymoma that is newly diagnosed or has come back. An MRI scan may be able to detect if and how far the tumor has spread more accurately than a standard computed tomography (CT) scan.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether thymoma staging by MRI is as accurate as staging by CT as compared to surgical staging.

SECONDARY OBJECTIVES:

I. To determine whether evaluation of phrenic nerve paralysis by functional MRI is as accurate as the fluoroscopic "sniff test" as compared to surgical evaluation of phrenic nerve involvement.

II. To determine whether fast novel MRI sequences are as accurate as conventional MRI sequences for staging thymoma, when comparing to surgical staging.

OUTLINE:

Patients undergo an MRI scan over 45-60 minutes and a diaphragm fluoroscopy 30 days before surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled to meet with a thoracic surgeon from MD Anderson Cancer Center (ACC) for resection of newly diagnosed thymoma or thymoma recurrence in the chest and scheduled for surgery

Exclusion Criteria:

* Children, defined as individuals younger than 18 years old on the preoperative visit with the thoracic surgeon
* Pregnant patients
* Patients unable to understand the consent form
* Patients with metal within the chest and pacemakers
* Patients with a known allergic reaction to gadolinium, who will have their MRI performed without contrast
* Patients with glomerular filtration rate (GFR) < 60 ml/min, who will have their MRI performed without contrast
* Patients with an allergy to iodinated contrast material will follow departmental routine policy, that is those with anaphylaxis will have their CT performed without intravenous contrast and others will be prepped as for departmental guidelines for routine chest CT
* Patients with abnormal renal function will have their CT study perform as per DI's iodinated contrast administration guidelines, and no contrast will be administered with GFR lower than 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06-08 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of magnetic resonance imaging (MRI) staging | Up to 10 years
  Will be compared to staging done by computed tomography (CT). McNemar's test will be used to compare the accuracy for the following five sets of comparisons: spin echo (SE) T1 compared versus (vs.) liver acquisition with volume acquisition (LAVA)+ in-phase (IP)/out-of-phase (OP), Dixon versus fast spin echo (FSE) T2, LAVA+IP/OP+Dixon vs. SET1+FSET2, LAVA+IP/OP+Dixon vs. computed tomography (CT) scan, and SET1+FSET2 vs. CT scan. A p value less than 0.05 will be defined as significant. A p value less than 0.05 will be defined as significant.

SECONDARY OUTCOMES:
Accuracy of phrenic nerve paralysis by functional MRI | Up to 10 years
  Will be evaluated against the fluoroscopic "sniff test" and compared to surgical evaluation of phrenic nerve involvement. The outcome is the binary indicator of whether the phrenic nerve is involved. The accuracy rate will be calculated for each of the three tested methods. And the method with the highest accuracy will be compared with the method with the medium accuracy and the method with least accuracy separately, using McNemar's test.
Accuracy of fast novel MRI sequences | Up to 10 years
  Will be evaluated against conventional MRI sequences for staging thymoma when compared to surgical staging. Will use the pathological stages as gold standard and calculate accuracy for the new shorter MRI sequences and current MRI sequences methods. Accuracy will be compared between two MRI techniques using McNemar's test. And the following five sets of comparisons will be tested: SE T1 compared vs. LAVA+ IP/OP, Dixon versus FSE T2, LAVA+IP/OP+Dixon vs. SET1+FSET2, LAVA+IP/OP+Dixon vs. CT scan, and SET1+FSET2 vs. CT scan. A p value less than 0.05 will be defined as significant.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Benveniste, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org